CLINICAL TRIAL: NCT01199484
Title: Specific Oral Tolerance Induction as an Useful Treatment in Two-year-old Children With Cow's Milk Allergy.
Brief Title: Specific Oral Tolerance Induction to Cow's Milk Allergy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General University Hospital of Valencia (Other)
Responsible Party: Antonio Martorell Aragones, Allergy Unit. University General Hospital
Organization: ValenciaUGH (Unknown)
Other Study IDs: SOTI-CMA
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Last update posted 2010-09-13 (Estimated); Status verified 2010-09

CONDITIONS: Food Hypersensitivity
Keywords: Cow's milk allergy; food allergy; oral desensitization; randomized trial; specific oral tolerance induction.
MeSH Terms: conditions — Food Hypersensitivity; Milk Hypersensitivity | interventions — Milk

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Cow's milk

SUMMARY:
Background: Limited published evidence shows specific oral tolerance induction (SOTI) to be a potential intervention option for cow's milk proteins (CMPs) allergy. Our hypothesis is that SOTI should be started early in order to improve its efficacy and prevent CMPs sensitization from evolving towards persistent allergy. The aim of this study was to evaluate the safety and efficacy of SOTI in 2-year-old children with cow's milk allergy, as a treatment alternative to elimination diet.

Methods: A total of 60 children between 24-36 months of age with IgE-mediated allergy to CMPs were included in this multicenter study and were randomly divided into two different groups. Thirty children (group A: treatment group) began SOTI immediately, whereas the remaining 30 (group B: control group) were kept on a milk-free diet and followed-up on for one year.

ELIGIBILITY:
Inclusion Criteria:

1. -Infants between 24-36 months of age.
2. -IgE-mediated allergy to CMPs meeting all the following diagnostic criteria:

   * Immediate-type clinical manifestations, skin (urticaria, angioedema and/or erythema), digestive (acute vomiting and/or diarrhea) or respiratory (bronchospasm and/or rhinitis) involvement in the first two hours after cow's milk ingestion.
   * Skin test readings ≥ 3 mm and specific IgE titers > 0.35 kU/l for whole cow's milk or someone of isolated CMPs (casein, alpha-lactalbumin, beta-lactoglobulin )
3. -Persistence of CMP allergy in the four weeks prior to tolerance induction, based on the following criteria:

   * Skin (prick) test readings ≥3 mm and specific IgE titers (CAP-FEIA) >0.35 kU/l for whole cow's milk or someone of isolated CMPs (casein, alpha-lactalbumin, beta-lactoglobulin )
   * Double-blind placebo-controlled challenge (DBPCFC) positive to cow's milk.
4. -Written informed consent from the parents.

Exclusion Criteria:

1. -Clinical manifestations of anaphylactic shock after the ingestion of cow's milk.
2. -Non-IgE-mediated or non-immunological adverse reactions to cow's milk.
3. -Malignant or immunopathological diseases and/or severe primary or secondary immune deficiencies.
4. -Patients receiving immunosuppressor therapy.
5. -Patients receiving beta-blockers (including topical formulations).
6. -Associated diseases contraindicating the use of adrenalin: cardiovascular disease or severe hypertension

Ages: 24 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child

CONTACTS AND LOCATIONS:
Locations (1):
- Allergy Unit. University General Hospital, Valencia, Valencia, Spain